CLINICAL TRIAL: NCT04859231
Title: Nutritive Effects of Cow's Milk-Based Formulas Through 18 Months of Age
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 6042
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Nutritive Effects on Brain Myelination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Other: Control
- Investigational (Experimental)
  Interventions: Other: Investigational
- Mother's-own Breast Milk (No Intervention)

INTERVENTIONS:
Other: Control — Cow's milk-based formula
  Arms: Control
Other: Investigational — Cow's milk-based formula with added source of enriched whey protein
  Arms: Investigational

SUMMARY:
This clinical trial will assess nutritive effects on brain myelination in infants assigned to receive one of two study formula or mother's own breast milk through 18 month's of age.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age)
* Birth weight of 2500 g (5 lbs 8 oz) or more
* Parent(s) or legal guardian agrees not to enroll infant in another interventional clinical study while participating in this study
* Signed informed consent obtained for infant's participation in the study
* Signed authorization obtained to use and/or disclose Protected Health Information for infant from birth through 18 months of age

Infants receiving formula:

* 3 to 60 days of age at randomization, inclusive (day of birth is considered day 0)
* Exclusively receiving infant formula for at least 72 hours prior to randomization
* Parent(s) or legal guardian has full intention to exclusively feed study formula during the study period

Infants receiving human milk:

* 150-180 days of age at registration, inclusive (day of birth is considered day 0)
* Mother has intention to predominately provide mother's own breast milk through at least 10 months of age

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* First degree relative with known autism, intellectual disability, schizophrenia, or bipolar disorder or an inherited disorder of myelination
* Major pre- and/or perinatal issues (such as maternal pre-eclampsia, placental abruption, maternal alcohol or illicit drug use during pregnancy)
* Major delivery complications (such as neonatal hypoxia or neonatal illness requiring a greater than 2-day NICU stay)
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as combined immunodeficiencies, DiGeorge syndrome, Wiskott-Aldrich syndrome, severe congenital neutropenia and secondary immunodeficiencies linked to HIV infection, Down syndrome or others)
* 5 minute APGAR < 7
* Infant was born large for gestational age (LGA) (as confirmed by the hospital birth records) from mother who was diabetic at childbirth
* Infant has been identified with inadequate weight gain or failure to thrive by a health care professional (HCP)
* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* Parent(s) or legal guardian unable to speak English at a level to provide informed consent

Infants receiving formula:

• Evidence of feeding difficulties or history of formula intolerance, such as vomiting or poor intake at time of randomization

Infants receiving human milk:

• Use of infant formula and/or donor milk more than three times per week prior to registration

Ages: 3 Days to 180 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
MR Imaging | 365 days of age
  Brain Imaging

SECONDARY OUTCOMES:
MR Imaging | 180 and 545 days of age
  Brain Imaging
Gap Overlap Paradigm | 180 and 365 days of age
Visual Expectation Paradigm | 180 and 365 days of age
A-not-B Task | 365 and 545 days of age
Bayley Scales of Infant and Toddler Development, Third Edition | 365 and 545 days of age
Body Weight | 180, 365 and 545 days of age
Length | 180, 365 and 545 days of age
Head Circumference | 180, 365 and 545 days of age
Recall of Study Feeding | 180, 275 (HM Reference group only), 365 and 545 days of age
  Feeding Questionnaire
Stool Microbiome Composition | 180, 365 and 545 days of age
  Sequence analysis using QIIME 2.0 (quantitative insights into microbial ecology)
Medically confirmed Adverse Events | Through study completion, on average 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831